CLINICAL TRIAL: NCT04709523
Title: Guided Bone Regeneration Using Bovine-derived Xenograft in Combination With or Without Injectable Platelet-rich Fibrin: a Randomized-controlled Clinical Trial
Brief Title: Guided Bone Regeneration Using Bovine-derived Xenograft in Combination With or Without Injectable Platelet-rich Fibrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gözde Işık, Lecturer, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ege Dentistry School
Record Dates: First submitted 2021-01-13; First posted 2021-01-14 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Bone Resorption
Keywords: Guided bone regeneration; Bovine-derived xenograft; Injectable platelet-rich fibrin
MeSH Terms: conditions — Bone Resorption | interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- i-PRF enriched bovine-derived xenograft (Experimental): Patients treated with i-PRF-enriched bovine-derived xenograft + resorbable membrane
  Interventions: Procedure: bovine-derived xenograft with i-PRF
- bovine-derived xenograft (Experimental): Patients treated with bovine-derived xenograft + resorbable membrane
  Interventions: Procedure: bovine-derived xenograft alone

INTERVENTIONS:
Procedure: bovine-derived xenograft with i-PRF — Bovine-derived xenograft was mixed with i-PRF and was placed in the augmentation site.
  Arms: i-PRF enriched bovine-derived xenograft
Procedure: bovine-derived xenograft alone — Bovine-derived xenograft was placed in the augmentation site.
  Arms: bovine-derived xenograft

SUMMARY:
The aim of the study was to compare the change in augmentation thickness after guided bone regeneration (GBR) using bovine-derived xenograft in combination with or without injectable platelet-rich fibrin (i-PRF).

This randomized-controlled clinical trial was conducted on patients with horizontal bone deficiency in the posterior regions of mandible. After implant placement, GBR procedures were randomly performed using i-PRF enriched bovine-derived xenograft (test group) or bovine derived xenograft alone (control group). Cone-beam computed tomography was taken at the implant sites immediately, and 6 months after surgery for assess the change in augmentation thickness as the primary outcome of the study. The secondary outcomes included marginal bone level and implant survival rate.

DETAILED DESCRIPTION:
The study was conducted on patients who had partially edentulism with horizontal deficiency of the alveolar bone in the posterior regions of mandible.

All patients were informed about treatment protocol of the study and also, the risks and benefits associated with participation. Each patient provided written informed consent prior to enrollment.

Randomization was performed after the dental implant surgeries and the patients were randomly assigned to one of the study groups:

Test group included 22 patients treated with GBR using i-PRF-enriched bovine-derived xenograft + resorbable membrane Control group included 22 patients treated with GBR using bovine-derived xenograft + resorbable membrane All patients underwent two-stage surgical protocol that performed by the same experienced surgeon. Following implant placement, i-PRF-enriched bovine-derived xenograft for the test group and bovine-derived xenograft alone for the control group was carefully positioned with light compression around the implants. Finally, the resorbable membrane was placed to cover the augmented area.

As the second stage of surgery, healing caps were placed and the implant-supported fixed prosthesis were completed in approximately one to two months.

ELIGIBILITY:
Inclusion Criteria:

* horizontal deficiency of the alveolar bone in the posterior regions of mandible
* absence of periodontal disease or previously treated
* with blood tests showing platelet counts at least 150.000 mm3
* ability to understand and accept the requirements of the study.

Exclusion Criteria:

* any disorders or infection at the implantation site or adjacent tissue
* tooth loss or extraction in the planned implant site within 6 months
* poor oral hygiene
* medical conditions that compromised tissue healing (uncontrolled diabetes, etc.)
* treatments with an interfering medications (bisphosphonates, steroids etc.)
* smoking habit
* pregnancy or nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-03-04 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Augmentation thickness | at immediately and at 6 months
  the change in augmentation thickness at surgical site.

SECONDARY OUTCOMES:
Marginal bone level | at immediately, at 6 months, at 12 months and at 24th months
  the change in marginal bone level around the implants after prosthetic loading